CLINICAL TRIAL: NCT00587470
Title: Angiotensin-II Blockade in Mitral Regurgitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Maurice Enriquez-Sarano M.D., Mayo Clinic Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1129-98; NCT00014846 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2010-10-15 (Estimated); Status verified 2010-10

CONDITIONS: Mitral Regurgitation
Keywords: valve, mitral, regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Atacand treatment.
  Interventions: Drug: Candesartan; Drug: atacand
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Candesartan — Maximum vasodilation.
  Other Names: atacand
  Arms: 1
Drug: atacand — maximum vasodilation
  Other Names: candesartan
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Mitral regurgitation (MR) is common in the elderly and its prevalence is increasing with the aging of the population. Organic MR, due to primary valvular lesions, initiates a cascade of complications determined by its degree. MR of severe degree is associated with excess mortality and high cardiac morbidity (heart failure, atrial fibrillation). It also causes left ventricular remodeling which induces left ventricular dysfunction, which in turn leads to poor clinical outcome. Surgery can eliminate MR, but carries immediate and long-term risks, especially in the elderly. Therefore, chronically decreasing the degree of MR is a major goal of medical therapy but such an effect is yet unproved because of conflicting results of small and mostly non-randomized series. Our recent preliminary studies suggest that a sustained decrease of degree of MR and improvement of left ventricular remodeling can be achieved with powerful reduction of afterload, obtained in particular with angiotensin-II receptor blockade. Therefore, the present proposal seeks to address gaps of knowledge regarding vasoactive treatment of MR through the verification of the following hypothesis: Hypothesis: Vasoactive therapy using angiotensin-II receptor blocker (Candesartan Cilexetil) weighed against placebo produces a sustained reduction of the consequences of organic MR. The specific aims are that the treatment a) decreases the degree of MR (decreases the regurgitant volume, primary end-point) and b) improves left ventricular remodeling (decreases the end-diastolic volume index, secondary end-point), as compared to placebo.

DETAILED DESCRIPTION:
Patients with MR organic (intrinsic valve disease), isolated (no other valve disease), moderate or more severe (regurgitant volume *30 mL/beat). A Clinical trial, randomized, placebo controlled, double-blind, without cross-over, of 1 year oral treatment with potent angiotensin-II receptor blockade using 32 mg Candesartan daily. The trial is preceded in all patients by an acute open-label study to determine tolerance and immediate response. The methods used to measure the end-points will be: a) Doppler-Echocardiography for quantitation of the degree of MR (measurement of regurgitant volume) using a combination of three simultaneous methods (quantitative Doppler, quantitative two-dimensional echocardiography, proximal flow convergence) and b) of left ventricular remodeling (end-diastolic volume index measured by echocardiography and by electron beam computed tomography). This single center study seeks to enroll a total of 90 patients. The analysis will be based on intention to treat and compare the regurgitant volume and left ventricular end-diastolic volume index measured after one year of treatment with the active drug or placebo. The results of the trial should provide strong evidence regarding medical treatment of patients with organic MR.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* 18 years old or older, with
* Mitral regurgitation on the basis of Color flow imaging
* Due to organic disease of the mitral valve on the basis of two-dimensional echocardiography
* Isolated (no valve disease other than functional tricuspid regurgitation on the basis of Doppler-Echocardiography)
* Pure (no mitral stenosis by Doppler echocardiography)
* Quantifiable by Doppler-Echocardiographic methods
* Of more than mild degree, defined as regurgitant volume * 30 mL/beat
* Occurring on native valves
* With Two-dimensional echocardiographic imaging allowing assessment of LV remodeling, and
* Asymptomatic (or mildly symptomatic but not considered as candidates for immediate surgery by their attending physician).

Exclusion Criteria:

* Associated aortic valve disease (more than trace aortic regurgitation by color flow imaging or mean gradient *25 mmHg)
* Associated mitral stenosis (mean gradient* 5 mmHg, valve area < 1.5 cm2)
* Associated congenital or pericardial diseases on the basis of Doppler echocardiography
* Intolerance to either AII blockers or Angiotensin converting enzyme inhibitors
* Intolerance to iodine contrast material
* Intolerance to intravenous echographic contrast agents
* Renal failure with creatinine * 2 mg/dl
* Blood pressure below 100 mmHg
* Known renal artery stenosis
* Ongoing therapy with hydralazine, calcium-entry blocking drugs or angiotensin converting enzyme inhibitors
* Known severe comorbidity such as liver disease, malignancy
* Pregnancy (A negative pregnancy test and effective contraceptive methods are required prior to enrollment of females of childbearing potential (not post-menopausal or surgically sterilized)), and
* Patients considered as requiring mitral valve surgery by their attending physician or with previous valve repair or replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1998-08; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Tolerance of the medication. | one year

SECONDARY OUTCOMES:
Decrease of severity of mitral regurgitation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maurice E. Sarano, M.D., Principal Investigator — Mayo Clinic Foundation
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States